CLINICAL TRIAL: NCT04279834
Title: Improving Outcomes for Patients With SDB and Insufficient Sleep
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Safwan Badr, Professor of Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1809001759; R01HL146059 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sleep Apnea; Insufficient Sleep Syndrome; Sleep; Hypertension
Keywords: Sleepiness; Hypertension; Sleep; Sleep Apnea; Endothelial Function; Alertness; Behavioral Intervention
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Deprivation; Hypertension; Sleepiness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAP Treatment (Active Comparator): Participants will receive a PAP device and will attend four weekly sessions to receive education about this treatment.
  Interventions: Behavioral: PAP Treatment
- Sleep Education I (Active Comparator): Participants will attend four weekly sessions to receive education about strategies to improve sleep.
  Interventions: Behavioral: Sleep Education I

INTERVENTIONS:
Behavioral: PAP Treatment — Motivational enhancement plus remote-monitoring and participant self-monitoring of PAP use.
  Arms: PAP Treatment
Behavioral: Sleep Education I — Motivational enhancement plus participant self-monitoring of sleep.
  Arms: Sleep Education I

SUMMARY:
The purpose of this study is to look at how sleep disordered breathing (SDB) and not getting enough sleep each night contribute to daytime sleepiness. The investigators also want to determine the treatment that works best for improving daytime sleepiness.

In this study, the investigators are comparing 2 programs that may improve symptoms of daytime sleepiness.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is associated with significant adverse health consequences including cardiovascular disease, motor vehicle accidents, daytime functional impairments, and mortality risk. A significant proportion of the populace has mild to moderate SDB.

This study is a randomized control trial (RCT) to test the efficacy of a program combining patient monitoring with behavioral techniques across Positive Airway Pressure (PAP) and sleep education. Screening for sleep apnea will be performed based on a phone screening questionnaire and an initial polysomnography (collected from another clinic or collected by research staff). Both objective (actigraphy, Psychomotor Vigilance Test, 24 hour blood pressure monitoring, office blood pressure, and EndoPATTM) and self-report (questionnaire/diary) sleep measures will be collected, as well as other health-related measures. Participants with an Apnea Hypopnea Index (AHI) between 5 and 30, and who meet all inclusion/exclusion criteria will be randomized to one of two educational programs.

Both groups will receive education about SDB and sleep, but only one group will receive PAP devices. This information will be provided to participants as part of the 4-session intervention. Follow-up assessments will be conducted immediately following the intervention and after 3-months.

Main study outcomes (lapses, daytime sleepiness, endothelial function and ambulatory blood pressure) will be assessed at baseline, post treatment and 3 month. Data will be analyzed using "intention to treat" principles, and appropriate statistical methods for clinical trials.

ELIGIBILITY:
Inclusion Criteria for enrollment are:

* Over age 18 years
* Diagnosed with mild to moderate sleep disordered breathing (SDB) (Apnea Hypopnea Index of 5-30)

Additional Inclusion Criteria for randomization will be:

* ESS score >6
* Total sleep time <7 hours at least 4 nights per week, based on baseline sleep diary.

Exclusion Criteria:

* Current use of PAP or oral appliance therapy for SDB
* Severe respiratory or cardiovascular disease (e.g., ventilatory failure, congestive heart failure)
* A recent health event that may affect sleep (e.g. recent surgery or hospitalization)
* Current alcohol or substance use disorder (<90 days sobriety) or significant unstable psychiatric comorbidity (e.g., suicidal ideation, psychosis)
* Pregnancy or within 6 months post-partum
* Commercial drivers and individuals at risk for motor vehicle accidents (MVA) or ESS>18
* Significant comorbid sleep disorders (e.g., severe insomnia, narcolepsy); and
* Central sleep apnea (defined as central apnea/hypopnea index >5, and >50% of total AHI).
* Use of sedative-hypnotic medications higher than the maximal acceptable therapeutic dose range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 3-months after randomization
  ESS is an 8-item questionnaire that assesses general level of daytime sleepiness. Total score ranges from 0 - 24, with higher scores indicating greater sleepiness.

SECONDARY OUTCOMES:
Reactive hyperemia index | 3-months after randomization
  Endothelial function will be measured by peripheral arterial tonometry (PAT) collected by fingertip sensor. Proprietary software is used to calculate a reactive hyperemia index.
24-hours Ambulatory Blood Pressure | 3-months after randomization
  Blood pressure will be monitored over a 24-hour period. Mean 24-hour blood pressure, mean daytime (rise time - bed time), and mean nocturnal (bed time - rise time) blood pressure will be calculated.
Fatigue Severity Scale (FSS) | 3-months after randomization
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Answers are scored on a point scale of 1 to 7 from strongly disagree to strongly agree. The minimum possible score is 9 and highest score is 63. A higher score indicates more severe fatigue and impact on the person's activities.
Psychomotor Vigilance Test (PVT) | 3-months after randomization
  PVT is a performance measure of alertness and vigilance. Reaction time to a visual cue, delivered at random intervals varying from 2 to 10 seconds, is measured. The total number of lapses (reaction time >500ms) during the 10 minute test will be used as a measure of objective alertness.

CONTACTS AND LOCATIONS:
Overall Officials: M. Safwan Badr, MD, MBA, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No